CLINICAL TRIAL: NCT03354546
Title: Creation, Evaluation and Validation of a Preoperative Frailty Index Using Health Administrative Data: a Population-based Cohort Study
Brief Title: Development and Validation of a Preoperative Frailty Index Using Health Administrative Data
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: DM8
Record Dates: First submitted 2017-11-17; First posted 2017-11-28 (Actual); Results first posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-05

CONDITIONS: Frail Elderly Syndrome; Surgery; Outcomes; Predictive Value of Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Elective noncardiac surgery: Individuals having major noncardiac surgery following an elective hospital admission
  Interventions: Diagnostic Test: Frailty index
- Emergency general surgery: Individuals having general surgery following an urgent hospital admission
  Interventions: Diagnostic Test: Frailty index

INTERVENTIONS:
Diagnostic Test: Frailty index — A frailty index composed of variables from health administrative data that cover multi-system health issues. Deficits will be coded as present or absent, and the number of deficits present will be divided by the total number of deficits present to provide an overall score between 0-1.

SUMMARY:
The investigators will create a frailty index using health administrative data available for older people having surgery. The index will be based on the Canadian Study of Health and Aging Frailty Index and standard recommendations for creation of frailty indices.

DETAILED DESCRIPTION:
The investigators will create a frailty index using health administrative data available for older people having surgery. The index will be based on the Canadian Study of Health and Aging Frailty Index and standard recommendations for creation of frailty indices.

Once derived the index will be tested to measure its association with outcomes, as well as its discrimination. Various representations of the frailty index will be tested (primary-as a continuous measure; secondary as a binary, categorical and fractional polynomial variable). Performance in subgroups will also be evaluated,

ELIGIBILITY:
Inclusion Criteria:

* Having elective or emergency noncardiac surgery

Exclusion Criteria:

* no provincial health insurance number

Min Age: 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All individuals 66 years of older on the day of their surgery
Sampling Method: Non-Probability Sample
Enrollment: 511285 (Actual)
Dates: Start 2002-04-01 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2016-03-31 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Elective: Individuals having major noncardiac surgery following an elective hospital admission
  Frailty index: A frailty index composed of variables from health administrative data that cover multi-system health issues. Deficits will be coded as present or absent, and the number of deficits present will be divided by the total number of deficits present to provide an overall score between 0-1.
- Emergency: Individuals having general surgery following an urgent hospital admission
  Frailty index: A frailty index composed of variables from health administrative data that cover multi-system health issues. Deficits will be coded as present or absent, and the number of deficits present will be divided by the total number of deficits present to provide an overall score between 0-1.
Period: Overall Study
Arm/Group | Elective | Emergency
Started | 415704 | 95581
Completed | 415704 | 95581
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Elective Surgery: Individuals having major noncardiac surgery following an elective hospital admission
  Frailty index: A frailty index composed of variables from health administrative data that cover multi-system health issues. Deficits will be coded as present or absent, and the number of deficits present will be divided by the total number of deficits present to provide an overall score between 0-1.
- Emergency Surgery: Individuals having general surgery following an urgent hospital admission
  Frailty index: A frailty index composed of variables from health administrative data that cover multi-system health issues. Deficits will be coded as present or absent, and the number of deficits present will be divided by the total number of deficits present to provide an overall score between 0-1.
- Total: Total of all reporting groups
Arm/Group | Elective Surgery | Emergency Surgery | Total
Number analyzed (Participants) | 415704 | 95581 | 511285
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Analysis for elective and emergency surgery groups were further separated into frail and not frail participants
  years
    Frail: number analyzed (Participants) | 119824 | 40038 | 159862
    Frail | 76 (6) | 76 (6) | 76 (6)
    Not Frail: number analyzed (Participants) | 295880 | 55543 | 351423
    Not Frail | 73 (6) | 73 (6) | 73 (6)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Analysis for elective and emergency surgery groups were further separated into frail and not frail participants
  Participants
    Frail: number analyzed (Participants) | 119824 | 40038 | 159862
    Frail: Female | 58953 | 21420 | 80373
    Frail: Male | 60871 | 18618 | 79489
    Not Frail: number analyzed (Participants) | 295880 | 55543 | 351423
    Not Frail: Female | 165693 | 30493 | 196186
    Not Frail: Male | 130187 | 25050 | 155237

OUTCOME MEASURES:

1. Primary Outcome: Survival for One Year After Surgery
Description: Still being alive (no death date) in the registered persons database Outcome is binary, exposure is per 0.1 unit increase
Time Frame: Date of surgery to 365 days after surgery
Population: We measured the unadjusted and adjusted associations between the pFI and postoperative outcomes in our elective surgery cohort. The unadjusted analysis contained only the pFI. Data was not collected from Emergency Surgery patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Elective Surgery | Emergency Surgery
Number analyzed (Participants) | 415704 | 0
Participants | 396164 | 0

2. Secondary Outcome: Institutional Discharge
Description: Discharge to long term care or continuing care facility at the time of hospital discharge
Time Frame: Date of surgery to date of hospital discharge, or up to one year after surgery (whichever comes first)
Population: We measured the unadjusted and adjusted associations between the pFI and postoperative outcomes in our elective surgery cohort. The unadjusted analysis contained only the pFI. Data not collected from Emergency Surgery patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Elective Surgery | Emergency Surgery
Number analyzed (Participants) | 415704 | 0
Participants | 57666 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: All-Cause Mortality was monitored
Arm/Group | Elective Noncardiac Surgery | Emergency General Surgery
All-Cause Mortality (participants affected / at risk) | 19540/415704 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Some variables underlying the pFI, such as pharmacy and home-support care data, may not be available in all data systems. Additionally, while the ACG system is the most widely used population-risk software in the world, it is not universally available, and diagnostic codes underlying its clusters are not openly disseminated. Our results represent associations, not causal relationships.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No